CLINICAL TRIAL: NCT05222906
Title: A Phase 3, Multicenter, Multinational, Randomized, Double-blind, Double-dummy, Active-comparator Study to Evaluate the Efficacy and Safety of Venglustat in Adult and Pediatric Patients With Gaucher Disease Type 3 (GD3) Who Have Reached Therapeutic Goals With Enzyme Replacement Therapy (ERT)
Brief Title: Study to Evaluate the Efficacy and Safety of Venglustat in Adult and Pediatric Patients With Gaucher Disease Type 3
Acronym: LEAP2MONO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17215; U1111-1265-6930 (Registry Identifier: ICTRP); 2024-514381-39 (Registry Identifier: CTIS); 2021-005402-10 (EudraCT Number)
Record Dates: First submitted 2022-01-20; First posted 2022-02-03 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Gaucher's Disease Type III
MeSH Terms: conditions — Gaucher Disease | interventions — venglustat; imiglucerase

STUDY DESIGN:
Intervention Model Description: Double Dummy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the open-label extended treatment period all participants will receive open label venglustat.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Venglustat (Experimental): Venglustat
  Interventions: Drug: Venglustat
- Cerezyme (Active Comparator): Cerezyme
  Interventions: Drug: imiglucerase

INTERVENTIONS:
Drug: Venglustat — tablet; oral
  Arms: Venglustat
Drug: imiglucerase — sterile lyophilized product; intravenous
  Other Names: Cerezyme®
  Arms: Cerezyme

SUMMARY:
This is a parallel arm, Phase 3, double-blind, double-dummy, active-comparator, 2 arm study to evaluate the efficacy and safety of daily oral venglustat versus intravenous Cerezyme infusions every two weeks for improvement or stabilization of the neurological manifestations and maintenance of systemic disease stability in participants aged ≥12 and <18 years and adult patients with Gaucher disease Type 3 (GD3) who have been treated with Enzyme Replacement Therapy (ERT) for at least 3 years.

DETAILED DESCRIPTION:
Screening period: 45 days

Double blind, double-dummy, primary analysis treatment period: 52 weeks

Open label extended treatment period: minimum of 52 weeks due to a common study end of treatment date

Follow up phone call: 30-37 days after end of treatment

ELIGIBILITY:
Inclusion Criteria:

* The participant has received ERT (Cerezyme or other ERT; as deemed appropriate by local regulations) for at least 3 years prior to enrollment, on a stable dose for at least 6 months, is deemed clinically stable for at least 1 year by the Investigator and is within the therapeutic goals as all of the following:

  * Hemoglobin level of ≥11.0 g/dL for females and ≥12.0 g/dL for males
  * Platelet count ≥100 000/mm3
  * Spleen volume <10 multiples of normal (MN)
  * Liver volume <1.5 MN
  * No bone crisis and free of symptomatic bone disease such as bone pain attributable to osteonecrosis and/or pathological fractures within 3 months prior to screening
* Adult participant is ≥18 years of age
* Pediatric participant is ≥12 years <18 years of age
* The participant has a clinical diagnosis of GD3 and a documented deficiency of acid beta-glucosidase activity confirming this diagnosis.
* The participant has a modified SARA score of 1 or above.
* The presence of gaze palsy, predominantly horizontal, with slow or absent saccades.
* If the participant has a history of seizures, they are well controlled under appropriate medication not identified as a strong or moderate inducer or inhibitor of CYP3A.
* Participants ≥ 30 kg of weight
* Contraception for sexually active male or female participants; not pregnant or breastfeeding; no sperm donating for male participant
* Signed written informed assent/consent

Exclusion Criteria:

* The participant is blood transfusion-dependent.
* Prior esophageal varices or liver infarction or current liver enzymes (alanine aminotransferase [ALT]/ aspartate aminotransferase [AST]) or total bilirubin >2 times the upper limit of normal, unless the participant has a diagnosis of Gilbert Syndrome.
* The participant has any clinically significant disease, other than GD, including cardiovascular (congenital cardiac defect, coronary artery disease, valve disease or left sided heart failure; clinically significant arrhythmias or conduction defect), hepatic, gastrointestinal, pulmonary, neurologic, endocrine, metabolic (eg, hypokalemia, hypomagnesemia) or psychiatric disease, other medical conditions, or serious intercurrent illnesses that may preclude participation in the opinion of the Investigator.
* The participant has renal insufficiency, as defined by an estimated glomerular filtration rate <30 mL/min/1.73m2 at the screening visit.
* The participant has a history of cancer, except for basal cell carcinoma.
* The participant has progressive myoclonic epilepsy.
* The participant is pregnant (has a positive serum beta-human chronic gonadotropin [β-hCG]) or lactating.
* The participant requires use of invasive ventilatory support.
* The participant requires use of noninvasive ventilator support while awake for longer than 12 hours daily.
* The participant is scheduled for in-patient hospitalization including elective surgery, during the study.
* The participant has had a major organ transplant (eg, bone marrow or liver).
* A history of drug and/or alcohol abuse within the past year prior to the screening visit.
* Chaperone therapy within 6 months, substrate reduction therapy other than venglustat within 6 months or venglustat substrate reduction therapy prior to enrollment.
* Exposure to any investigational drug within the last 30 days or 5 half-lives from screening, whichever is longer.
* The participant has received strong or moderate inducers or inhibitors of CYP3A within 14 days or 5 half-lives from screening, whichever is longer, prior to screening. This also includes the consumption of grapefruit, grapefruit juice, or grapefruit containing products within 72 hours of starting venglustat. The participant is unwilling to abstain from consumption of grapefruit, grapefruit juice, or grapefruit containing products for the duration of the treatment period.
* The participant, in the opinion of the investigator, is unable to adhere to the requirements of the study or unable to undergo study assessments (eg, contraindication for MRI).
* Type of participant and disease characteristic: the participant has had a total splenectomy prior to enrollment. The patient had a partial splenectomy within 3 years prior to randomization.
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in Scale for Assessment and Rating of Ataxia (SARA) modified total score | From baseline to Week 52
Change in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) total scale index score | From baseline to Week 52

SECONDARY OUTCOMES:
Percent change in spleen volume | From baseline to Week 52
Percent change in liver volume | From baseline to Week 52
Change in hemoglobin level | From baseline to Week 52
Percent change in platelet count | From baseline to Week 52
Percent change in CSF GL-1 and lyso-GL-1 levels | From baseline to Week 52
Percent change in plasma GL-1 and lyso-GL-1 levels | From baseline to Week 52
Number of patients with treatment emergent adverse events (TEAEs)/ serious adverse events (SAEs)/ adverse events of special interest (AESIs) | From baseline to max of 4.5 years
Change in score of Beck Depression Inventory II (BDI-II) during the treatment-emergent period (for participants 13 years of age and above at baseline) | From baseline to Week 52
Change in Patient Health Questionnaire 9 (PHQ-9) during the treatment-emergent period (for participants 12 years of age at baseline) | From baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (22):
- United States (4):
  - Yale University School of Medicine - Investigational Site Number: 8400003, New Haven, Connecticut
  - University of Iowa - Investigational Site Number: 8400002, Iowa City, Iowa
  - Texas Oncology - Medical City Dallas Site Number : 8400008, Dallas, Texas
  - Lysosomal & Rare Disorders Research & Treatment Center, Inc - Investigational Site Number: 8400001, Fairfax, Virginia
- Hospital de Ninos - Investigational Site Number: 320001, Buenos Aires, Argentina
- Children's Hospital Research Institute of Manitoba - Investigational Site Number: 1240001, Winnipeg, Manitoba, Canada
- China (4):
  - National Taiwan University Hospital-Investigational Site Number: 1580001, Taipei, Taiwan
  - Peking Union Medical College Hospital - Investigational Site Number: 1560001, Beijing
  - The First Affiliated Hospital - Investigational Site Number: 1560002, Guangzhou
  - Xinhua Hospital - Investigational Site Number: 1560004, Shanghai
- France (2):
  - 47-87, boulevard de l'hôpital - Investigational Site Number: 2500003, Paris
  - Hopital Necker - Investigational Site Number: 2500001, Paris
- SphinCS GmbH - Investigational Site Number: 2760001, Hochheim am Main, Germany
- Debreceni Egyetem, Klinikai Központ, Reumatológiai Klinika - Investigational Site Number: 3480001, Debrecen, Hungary
- Italy (2):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Investigational Site Number : 3800003, Milan, Lombardy
  - Azienda Ospedaliera Universitaria (AOU) "Federico II" - Investigational Site Number: 3800002, Napoli
- Japan (2):
  - Odawara Municipal Hospital-Investigational Site Number : 3920002, Odawara, Kanagawa
  - Tohoku University School of Medicine - Investigational Site Number: 3920001, Sendai
- Turkey (Türkiye) (3):
  - Cukurova University Medical School Hospital-Investigational Site Number : 7920001, Adana
  - Gazi University Medical Hospital-Investigational Site Number : 7920002, Ankara
  - Istanbul University Medical Faculty Hospital-Investigational Site Number : 7920004, Istanbul
- Investigational Site Number : 8260001, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17215 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25262&tenant=MT_SNY_9011